CLINICAL TRIAL: NCT05135702
Title: Effect of Propionic Acid Supplementation on Endothelial Function in Patients With Coronary Artery Disease
Brief Title: Effect of Propionic Acid Supplementation on Endothelial Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Michael E. Widlansky, Professor of Medicine and Pharmacology, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PRO39540
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases; Endothelial Dysfunction
MeSH Terms: conditions — Cardiovascular Diseases | interventions — sodium propionate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium Propionate First (Experimental): Subjects in this arm will consume 500mg sodium propionate powder twice daily for four weeks, mixed into their food/drink. This is followed by four weeks of placebo twice daily.
  Interventions: Dietary Supplement: Sodium Propionate; Dietary Supplement: Placebo
- Placebo First (Placebo Comparator): Subjects in this arm will consume a placebo twice daily for four weeks, mixed into their food/drink. This is followed by four weeks of 500mg sodium propionate powder, twice daily.
  Interventions: Dietary Supplement: Sodium Propionate; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sodium Propionate — a 500 mg powder dietary supplement that can be mixed into food or drinks. It will be taken twice daily for four weeks.
Dietary Supplement: Placebo — a color, size, calorie, and consistency-matched powder dietary supplement that can be mixed into food or drinks. It will be taken twice daily for four weeks.

SUMMARY:
Coronary Artery Disease (CAD) remains a leading cause of morbidity and mortality worldwide despite improved mitigation of traditional risk factors. Large association studies have linked the gut microbiome alterations with inflammation, CAD, and traditional CAD risk factors. Subsequent studies have shown concomitant improvements in gut dysbiosis, inflammation, and cardiometabolic diseases using probiotics and other gut-modulating therapies. To date, many studies have shown a correlative relationship between intestinal bacteria composition and the presence of CAD, or severity of heart attacks, but few have begun to elucidate potential metabolic and immunologic mechanisms.

The investigator's recently supplemented Lactobacillus plantarum 299v in men with stable CAD, which improved systemic inflammation and brachial artery flow-mediated dilation (BA-FMD) - a measure of endothelial function and a predictive CAD precursor. Improvement in BA-FMD positively correlated with increased serum propionic acid (PA) concentrations. PA is a gut microbiome-derived short chain fatty acid (SCFA) with known human vascular receptors and implicated in endothelial function, innate immunity, and glucose homeostasis.

Whether PA is mediating improvement in endothelial dysfunction or inflammation in the investigator's prior experiment remains unknown. The investigator's objective is to determine whether endothelial cell function is improved by dietary supplementation of sodium propionate in patients with established coronary artery disease. Furthermore, the investigators wish to elucidate to what extent inflammation is reduced by this therapy, by both measuring serum inflammatory markers and by seeing if plasma from treated patients induces anti-inflammatory transcriptomic responses from cultured endothelial cells and peripheral blood mononuclear cells, both of which are involved in atherosclerosis.

Specific Aim 1 will determine the impact of dietary PA supplementation on endothelial function and traditional CAD risk factors in patients with CAD. The investigators will utilize ultrasound to assess the percent change in BA-FMD before and after dietary PA supplementation. The extent of endothelium-dependency of these responses will be tested by measuring BA-FMD following nitroglycerin administration. The investigators will also measure markers representative of traditional CAD risk factors, such as lipid levels and HgbA1C.

Specific Aim 2 will determine anti-inflammatory changes in vivo and in transcriptomic signatures of cultured EC and PBMCs induced by dietary PA. The investigators will measure changes to systemic serum inflammatory markers involved in atherosclerotic processes using a targeted metabolomics approach, using plasma from the investigator's cohort before and after PA supplementation. Plasma samples will be used to incubate aforementioned cells to compare transcriptomic signatures of cells subjected to pre-supplementation plasma versus post-supplementation plasma. The investigators will use Ingenuity Pathway Analysis to determine changes to inflammatory pathways and i.i.com to determine whether more anti-inflammatory signatures were induced.

Specific Aim 3 will determine the impact of PA supplementation on gut microbiome taxonomy and diversity. As an optional additional clinical study activity, the investigators will collect stool samples before and after dietary PA supplementation, subject samples to multiplex 16S RNA sequencing, and calculate the Shannon Diversity Index. This will help us determine changes in individual gut microbiome constituents and diversity of the entire population.

DETAILED DESCRIPTION:
Endothelial dysfunction (ED) is a pathological state of vessel function characterized by increased expression of pro-vasoconstrictive mediators and increased thrombotic risk. ED is associated with the development of atherosclerosis, including coronary artery disease (CAD), and with increased risk of cardiovascular events Therefore, there is an ongoing research effort to restore endothelial function in order to reduce the risk of cardiovascular morbidity associated with endothelial dysfunction.

The gut microbiome has been well correlated with the presence of CAD and alterations to the gut microbiome have been mechanistically linked to the severity of myocardial infarction. Animal experiments showed that alteration of gut bacteria with supplementation of Lactobacillus plantarum 299v (Lp299v) and vancomycin is associated with reduced leptin levels, size of myocardial infarction and improved post -ischemic cardiac function. In humans, dietary supplementation with Lp299v was associated with significant reductions in LDL-cholesterol, fibrinogen, and leptin concentrations in smokers.The investigatorsrecently showed in men with stable CAD that six weeks' supplementation with Lp299v improved endothelial function as assessed by brachial artery flow-mediated dilation (BA-FMD), a widely accepted noninvasive modality of assessing vascular endothelial function. This intervention concurrently reduced serum inflammatory markers IL-8, IL-12 and leptin, and post-probiotic plasma drove an anti-inflammatory transcriptomic response in cultured peripheral blood mononuclear cells. Interestingly, these beneficial changes were not accompanied by changes in gut microbiome constituents. Instead, the increase seen in BA-FMD was positively correlated with an increase in serum propionic acid, one of the short-chain fatty acids, a set of molecules produced by gut microbes and freely absorbed into human circulation. Propionic acid is known to improve endothelial function, reduce systemic inflammation, and improve glucose homeostasis in several models. These experiments suggested that Lp299v's beneficial effects were mediated by changes to the existing gut microbiome's metabolism as opposed to changes to microbial constituents. The investigators identified propionic acid as a potential mediator of these beneficial outcomes.

In this study, the investigator's objective is to assess if there is any impact of sodium propionate dietary supplementation on vascular endothelial function and on the levels of circulating inflammatory markers related to endothelial dysfunction. In addition, the investigators also will study if the impact on endothelial function is associated with either: anti-inflammatory changes in relevant vascular cell types (e.g. endothelial cells, peripheral blood mononuclear cells), or on the constituents of the gut microbiome itself.

Endothelial function is easily measurable by non-invasive means. Endothelial dysfunction measured non-invasively independently predicts future cardiovascular risk in patients both with and without clinically apparent cardiovascular disease. Conduit vessel endothelial function in humans is commonly quantified by measurement of BA-FMD, which represents the endothelium-dependent relaxation of a conduit artery-typically the brachial artery - due to an increased blood flow. BA-FMD correlates with impaired endothelium-dependent relaxation in the coronary arteries and is a commonly recognized "barometer" of cardiovascular risk. BA-FMD is an ideal surrogate marker of cardiovascular risk to monitor the acute impact of Lp299v supplementation on vascular endothelial function.

ELIGIBILITY:
Inclusion Criteria:

History of known coronary artery disease as defined by having one or more of the following:

* history of myocardial infarction
* angiogram demonstrative >=50% stenosis in at least 1 major epicardial coronary artery
* a previous stress test that showed evidence of ischemia (that has not been revealed to be a false positive test by angiography)
* CT coronary study showing EITHER a coronary artery calcium (CAC) score of >400, OR a description of "significant stenosis" of one or more epicardial arteries.

Exclusion Criteria:

1. Unstable angina or myocardial infarction by history, ECG, and/or enzymatic criteria within 1 month of enrollment.
2. LV dysfunction as defined by an LV ejection fraction documented as < 45% within 1 year of enrollment by an echocardiogram, MRI, or nuclear imaging.
3. Uncontrolled hypertension with a blood pressure greater than 170/100 mmHg at the screening visit.
4. Known history of chronic renal insufficiency, liver dysfunction, or cancer besides non-melanoma skin carcinomas or localized prostate cancer requiring systemic treatment within five years of enrollment.
5. Known history of cognitive impairment or inability to follow study procedures.
6. Patient with GI tract illness such as short gut syndrome, inflammatory bowel disease, or an ileostomy.
7. Patient with an implanted defibrillator or permanent pacemaker on which the potential participant is known to rely upon for greater than 50% of ventricular depolarizations.
8. Patients who received probiotics, prebiotics, or short chain fatty acid supplements (e.g. propionate, butyrate, acetate-containing supplements) within the past 4 weeks.
9. Patients who received antibiotics in the last 12 weeks.
10. Patients with dosing changes of vasoactive medications and HMG-CoA reductase inhibitors in the 6 weeks prior to enrollment.
11. Pregnancy
12. Those who are daily drinkers or use illicit drugs.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2027-07 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in baseline flow mediated dilation (FMD) at 4 weeks | baseline and week 4
  This is a measurement of endothelial function in the brachial artery

IPD SHARING:
Plan to Share IPD: Undecided